CLINICAL TRIAL: NCT02609789
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study in Healthy Subjects and Multiple Dose Study of JNJ-55920839 in Subjects With Mild to Moderate Systemic Lupus Erythematosus
Brief Title: A Single Ascending Dose Study in Healthy Participants and Multiple Dose Study of JNJ-55920839 in Participants With Mild to Moderate Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108073; 55920839SLE1001 (Other: Janssen Research & Development, LLC); 2014-005605-21 (EudraCT Number)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus; Healthy
Keywords: Systemic Lupus Erythematosus; JNJ-55920839; Healthy Volunteers; CNTO 6358
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — JNJ-55920839

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: Dose 1 (Experimental): Drug JNJ-55920839 or Placebo administered IV infusion Dose 1.
  Interventions: Drug: JNJ-55920839; Drug: Placebo
- Part A: Dose 2 (Experimental): Drug JNJ-55920839 or Placebo administered IV infusion Dose 2.
  Interventions: Drug: JNJ-55920839; Drug: Placebo
- Part A: Dose 3 (Experimental): Drug JNJ-55920839 or Placebo administered IV infusion Dose 3.
  Interventions: Drug: JNJ-55920839; Drug: Placebo
- Part A: Dose 4 (Experimental): Drug JNJ-55920839 or Placebo administered IV infusion Dose 4.
  Interventions: Drug: JNJ-55920839; Drug: Placebo
- Part A: Dose 5 (Experimental): Drug JNJ-55920839 or Placebo administered IV infusion Dose 5.
  Interventions: Drug: JNJ-55920839; Drug: Placebo
- Part A: Dose 6 (Experimental): Drug JNJ-55920839 or Placebo subcutaneous injection Dose 6.
  Interventions: Drug: JNJ-55920839; Drug: Placebo
- Part B (Experimental): Participants will receive 6 doses of JNJ-55920839 or placebo (every 2 weeks) as an IV infusion.
  Interventions: Drug: JNJ-55920839; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-55920839 — JNJ-55920839 will be administered as either IV infusion or subcutaneous injection.
  Other Names: CNTO 6358
Drug: Placebo — 0.9 percent (%) normal saline.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of JNJ-55920839 following single ascending intravenous (IV) dose administration in healthy participants and a single subcutaneous dose in healthy participants and multiple IV dose administrations in participants with mild to moderate Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase 1, randomized, placebo-controlled, multicenter study of JNJ-55920839. The study consists of Screening Period of 28 days. The healthy participants will have a 6-day/5-night inpatient period. All Participants will receive study agent on Day 1 and SLE Participants will receive additional doses on Days 15, 29, 43, 57, and 71. The total duration of participation for each participant will be approximately 13 weeks for healthy participants, 22 weeks for participants with SLE. All eligible participants will be randomly assigned to receive active agent or placebo. The study will be conducted in 2 parts. In Part 1, single ascending doses of JNJ55920839 or placebo will be administered to sequential cohorts of healthy participants as an IV infusion or as a subcutaneous injection. In Part 2, multiple doses of JNJ-55920839 or placebo will be administered as IV infusions to participants with SLE. Blood samples will be collected for assessment of pharmacokinetic and pharmacodynamics parameters in both part 1 and 2, along with assessment of safety and clinical outcomes. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Part A (Healthy Participants)

* Participant must be willing/able to adhere to the study visit schedule and other requirements, prohibitions, and restrictions specified in this protocol
* Participant must have a body weight in the range of 50 to 90 kilogram (kg), inclusive, and have a body mass index (BMI) of 18 to 30 kilogram per square meters kg/m^2, inclusive, at screening
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. The determination that there is no evidence of active underlying illness by physical examination must be recorded in the Participant's source documents and initialed by the investigator
* Participant must be healthy on the basis of clinical laboratory tests performed at screening
* Before randomization, a woman must be: Not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 international units per liters (IU/L) or mIU/mL); permanently sterilized (e.g., bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 4 months (>= 5 half-lives) after receiving last dose of study agent
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 4 months (>=5 half-lives) after receiving the last dose of study agent

Part B (Participants with Systemic Lupus Erythematosus)

* Participant must be willing/able to adhere to the study visit schedule and other requirements, prohibitions, and restrictions specified in this protocol
* Participant must have a body weight in the range of 40 to 100 kg, inclusive, and have a BMI of 18 to 30 kilograms per square meters (kg/m^2), inclusive, at screening
* Must meet Systemic Lupus International Collaborating Clinics (SLICC) criteria for diagnosis of lupus

Exclusion Criteria:

Part A (Healthy Participants)

* Coexisting medical conditions or past medical history: Participant currently has or has had a history of any clinically significant medical illness or medical disorders the investigator considers significant should exclude the participant, including (but not limited to), neuromuscular disorder, hematological disease, immune deficiency states, respiratory disease, cardiovascular disease (including poor peripheral venous access), hepatic or gastrointestinal (GI) disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease. Careful consideration should be given to whether the participant has had severe, progressive, or uncontrolled hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic/ cerebral, or psychiatric disease, or current signs and symptoms thereof
* Participant has a condition that might confound assessments including major surgery, substance abuse or acute illness
* Participant is a woman of childbearing potential or a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 4 months (>=5 half-lives) after the last dose of study agent

Part B (Systemic Lupus Erythematosus [SLE] )

* Participant with history or suspected occurrence of drug-induced SLE
* Participant has active Central nervous system (CNS) lupus or history of severe CNS lupus including but not limited to seizures, psychosis, transverse myelitis, CNS vasculitis and optic neuritis
* Participant currently has or has had a history of any clinically significant medical illness or medical disorders the investigator considers significant should exclude the Participant, including (but not limited to), neuromuscular disorder, hematological disease, immune deficiency states, respiratory disease, cardiovascular disease (including poor peripheral venous access), hepatic or gastrointestinal (GI) disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease. Careful consideration should be given to whether the Participant has had severe, progressive, or uncontrolled hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic/ cerebral, or psychiatric disease, or current signs and symptoms thereof
* Participant has had major surgery, (e.g., requiring general anesthesia) within 4 months before screening, or will not have fully recovered from surgery, or has surgery planned within 4 weeks prior to study agent administration or during the time the Participant is expected to participate in the study, or within 4 months (>=5 half-lives) after the last dose of study agent administration
* Participant has laboratory findings or biopsy results consistent with severe lupus nephritis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability of JNJ-55920839 (Part 1) | Through Week 13
  The incidence of TEAEs from treatment until the last scheduled follow-up visit will be summarized by treatment group.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability of JNJ-55920839 (Part 2) | Through Week 22
  The incidence of TEAEs from treatment until the last scheduled follow-up visit will be summarized by treatment group.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) after IV infusion in Part A | Up to Day 64 after dose
Maximum Observed Serum Concentration (Cmax) after SC injection in Part A | Up to Day 64 after dose
Maximum Observed Serum Concentration during a dosing interval (Cmax) after IV infusion in Part B | Up to Day 130 after dose
Area under the serum concentration versus time curve from time 0 to the time corresponding to the last quantifiable serum concentration (AUC0-t) after IV infusion in Part A | Up to Day 64 after dose
Area under the serum concentration versus time curve from time 0 to the time corresponding to the last quantifiable serum concentration (AUC0-t) after SC injection in Part A | Up to Day 64 after dose
Area under the serum concentration versus time curve between 2 defined sample points, t1 and t2 (AUCt1-t2) after IV infusion in Part B | Up to Day 130 after dose
Terminal half-life (T1/2) after IV infusion in Part A | Up to Day 64 after dose
Terminal half-life (T1/2) after SC injection in Part A | Up to Day 64 after dose
Terminal half-life (T1/2) after IV infusion in Part B | Up to Day 130 after dose
Bioavailability (F) after SC injection in Part A | Up to Day 64 after dose
Number of Participants With Antibodies to JNJ-55920839 after IV infusion in Part A | Up to Day 64 after dose
Number of Participants With Antibodies to JNJ-55920839 after SC injection in Part A | Up to Day 64 after dose
Number of Participants With Antibodies to JNJ-55920839 after IV infusion in Part B | Up to Day 130 after dose

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (16):
- United States (3):
  - Birmingham, Alabama
  - Rochester, Minnesota
  - Durham, North Carolina
- Belgium (2):
  - Leuven
  - Merksem
- Chisinau, Moldova
- Poland (2):
  - Otwock
  - Szczecin
- Romania (2):
  - Bucharest
  - Timișoara
- Spain (4):
  - Barcelona
  - Madrid
  - Santiago de Compostela
  - Seville
- Taiwan (2):
  - Kaohsiung City
  - Taichung

REFERENCES:
- [Derived] Jordan J, Benson J, Chatham WW, Furie RA, Stohl W, Wei JC, Marciniak S, Yao Z, Srivastava B, Schreiter J, Cesaroni M, Orillion A, Seridi L, Chevrier M. First-in-Human study of JNJ-55920839 in healthy volunteers and patients with systemic lupus erythematosus: a randomised placebo-controlled phase 1 trial. Lancet Rheumatol. 2020 Oct;2(10):e613-e622. doi: 10.1016/S2665-9913(20)30223-X. Epub 2020 Aug 21. PMID 38273624
- [Derived] Yao Z, Loggia L, Fink D, Chevrier M, Marciniak S, Sharma A, Xu Z. Pharmacokinetics and Pharmacodynamics of JNJ-55920839, an Antibody Targeting Interferon alpha/omega, in Healthy Subjects and Subjects with Mild-to-Moderate Systemic Lupus Erythematosus. Clin Drug Investig. 2020 Dec;40(12):1127-1136. doi: 10.1007/s40261-020-00978-4. Epub 2020 Oct 21. PMID 33085033